CLINICAL TRIAL: NCT03562936
Title: Prospective Observational Cohort Study of Patients With Symptomatic Degenerative Spinal Stenosis With and Without Degenerative Spondylolisthesis Not Scheduled for Surgery
Brief Title: The NORDSTEN Studies/The Observational Cohort Study
Acronym: NORDSTEN/OS
Status: Active, not recruiting | Type: Observational
Sponsor: Haukeland University Hospital (Other)
Collaborators: Møre og Romsdal Hospital Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 2011/2034-2
Record Dates: First submitted 2018-05-31; First posted 2018-06-20 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-08

CONDITIONS: Degenerative Lumbar Spinal Stenosis; Degenerative Spondylolisthesis
Keywords: LSS,DS

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The NORDSTEN- OS(Observational study) aim to study the natural course in patients with mild to moderate symptomatic lumbar spinal stenosis with and without degenerative spondylolisthesis. 10 years follow-up is planned.

The NORDSTEN-OS is one of three studies in The NORwegian Degenerative Spondylolisthesis and Spinal STENosis studies.

The two other studies are:

NORDSTEN-SST (Spinal stenosis trial) (NCT02007083); a randomized controlled trial comparing the clinical and radiological results in three different decompression techniques in patients with lumbar spinal stenosis. The NORDSTEN-DS (Degenerative spondylolisthesis) (NCT02051374); a randomized controlled trial comparing the outcome of surgery with decompression without fixation and decompression with fixation in patients with lumbar spinal stenosis and concurrent degenerative spondylolisthesis.

DETAILED DESCRIPTION:
Objectives:

1. A longitudinal observation of clinical- and radiological development with 5- and 10 years follow-up. Variables predicting clinical deterioration or improvement, and outcome measurements including time from inclusion to time for surgery, will be analyzed. We will use predictive models appropriate to the type of data each prognostic outcome measure represents. For example the repeated pain and disability measures will be analysed using linear mixed models. Logistic regression models with no more than 1 variable per 10 events will be used to analyse associations between prognostic factors and disability. Multivariate analysis will identify the predictive prognostic factors in the demographic, physical, social and radiological domains. The number of factors that will be entered in the multivariate analysis will be condensed by univariate pre-testing and omitting highly correlated factors. The prognostic value of both single and combined variables will be addressed by calculating sensitivity, specificity, positive and negative likelihood ratios in a standard way.

   Time to surgery will be modeled using Kaplan-Meier plot. Depending on number of treated patients the effect of selected covariates on time to surgery will be evaluated using the Cox model.
2. 1) To investigate differences between patients in the observational cohort and patients treated surgically in NORDSTEN-SST and NORDSTEN-DS, by comparing baseline demographic-, clinical-, and radiological data. Patients in the NORDSTEN-OS with lumbar spinal stenosis and a verified degenerative spondylolisthesis of ≥ 3mm will be compared to patients in the NORDSTEN-DS. Patients in the NORDSTEN-OS with lumbar spinal stenosis without degenerative spondylolisthesis will be compared to patients in the NORDSTEN-SST. We will use descriptive statistics to compare the patient groups. For each of the variables we will compare measures of central tendency such as mean and median, and measures of variability such as variance and quantiles. We will also plot distributions of certain variables using histograms or fitted densities, in order to easier compare and see similarities and differences between the groups.

Baseline data Demographical data: Age, gender, BMI, education and native language. Status regarding: marriage, smoking, work and disability benefits.

Clinical data: duration of symptoms (back pain and leg pain) and use of analgetics, Patient reported outcome measures: Oswestry Disability Index (ODI 2.0), Zurich Claudication Questionnaire, EQ-5D and Numeric Rating Scale for leg pain and back pain. Hopkins symptom check list (HSCL-25) HSCL-25 is a PROM for assessment of psychological variables. It covers emotional distress, scores range from 1 to 4, with lower scores indicating less severe symptoms.

Radiological data: Standing x-rays; anterior-posterior (AP), lateral and functional images (lateral- extension and flexion) and MRI.

Radiological evaluations Standing x-ray with functional images and MRI will be performed at baseline-, 5-, and 10 years follow-up. Additionally, patients with lumbar spinal stenosis and concomitant degenerative spondylolisthesis at baseline undergo functional radiographs at 2 years follow-up. One musculoskeletal radiologist and two surgeons (Orthopedic surgeon and Neurosurgeon) will perform the radiological interpretations using Picture Archiving and Communication System (PACS), Sectra, Sweden.

MRI of the lumbar spine, including T1 and T2 sequences in the axial and sagittal planes. The following variables will be measured:

Measurements quantifying the degree of stenosis:

Morphologic grading according to the method described by Schizas et al. The grading is based on the cerebrospinal fluid/rootlet ratio, and is scaled from A-D, where A is no stenosis, B moderate stenosis, C severe stenosis and D extreme stenosis.

Measurements from sagittal plane T1 MRI sequences for grading of foraminal stenosis using the method of Lee et al.

The presence or absence of redundant nerve root sign.

Measurements when degenerative spondylolisthesis is present:

Measurement of the facet joint orientation will be done by MRI images in the transverse plan using the method of Berleman et al.

Degree of disc degeneration according to Pfirrmann et al and Modic et al. Qualitative measurement of facet joint fluid.

Qualitative measurement of disc height.

Skeletal x-rays:Standard images; frontal and lateral view of L1 to S1 in standing position.Extension- and flexion images; lateral view of L1 to S1 with respectively maximal flexion and maximal extension.

Measurement of lumbar lordosis (L1-S1),sacral slope Measurements from the radiographs for calculating vertebral sagittal olisthesis and segmental instability will use the method of Dupuis et al.

ELIGIBILITY:
Inclusion Criteria:

* Presence of clinical symptoms of spinal stenosis. Neurogenic claudication or radiating pain to one or both lower limbs
* Radiological findings corresponding to the clinical symptoms of LSS. Central stenosis or lateral recess stenosis with or without degenerative spondylolisthesis
* Able to understand Norwegian language, both spoken and written
* Able to give informed consent and to answer the questionnaires
* Over 18 years of age

Exclusion Criteria:

* Not willing to give written consent
* Participation in other clinical trial that may interfere with this trial
* American Society of Anesthesiologists (ASA) 4 or 5
* Age older than 80 years
* Not able to comply fully with the protocol, including treatment, follow-up or study procedures (psychosocially, mentally and physically)
* Presence of cauda equina syndrome (bowel and bladder dysfunction) or complete motor deficit
* Presence of an isthmic defect in pars interarticularis
* Former fracture of the thoracolumbar region
* Previous surgery in the lumbar region
* Distinct symptoms in one or both legs due to other diseases, e.g. polyneuropathy, vascular claudication or osteoarthritis
* Lumbosacral scoliosis of more than 20 degrees verified on standing x-ray AP-view

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with symptomatic LSS with and without LDS referred to the participating orthopedic- or neurosurgical departments will be eligible for inclusion in the observational cohort. The burden of symptoms is considered not to be severe enough to opt for surgical treatment, and this conclusion is made through informed shared decision-making between surgeon and patient. Patients will be given verbal and written information about this observational study. If willing to participate, the patients sign an informed consent. The treatment of these patients will be pragmatic "usual care". There will not be any planned specific conservative treatment, but the surgeon can recommend specific conservative treatments in any case if preferred
Sampling Method: Non-Probability Sample
Enrollment: 284 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Oswestry Disability Index (ODI) version 2.0 | Baseline and follow-up at 2,5 and 10 years
  ODI is a patient reported outcome measure (PROM) comprising 10 sections where the patient is supposed to mark the most appropriate item. ODI scores range from 0 to 100, with higher score indicating more severe pain and disability. ODI is recommended by international expert panels for the evaluation of disability in clinical trials and commonly used by physicians treating patients with back-related symptoms. It has been translated and validated for applications with Norwegian patients. The change in ODI from baseline to follow-up will be registered.

SECONDARY OUTCOMES:
Zürich Claudication Questionnaire (ZCQ) | Baseline and follow-up at 2,5 and 10 years
  A PROM evaluating disorder-specific functional capacity covering three domains: symptom severity (score 1-5), physical function (score 1-4), and patient satisfaction (Score 1-4) The change in ZCQ from baseline to follow-up will be registered
Numeric Rating Scale (NRS) for back and leg pain. | Baseline. Follow-up at 2,5 and 10 years
  NRS is a PROM that assesses self-reported pain from 0 (no pain) to 10 (the worst pain imaginable). The change in NRS for back- and leg pain from baseline to follow-up will be registered.
EuroQol 5 dimensions questionnaire (EQ-5D). | Baseline and follow-up at 2,5 and 10 years
  EQ-5D is a generic PROM for the evaluation of quality of life comprising 5 questions relating to mobility, self-care, usual activity, pain/discomfort, and anxiety/depression. Each question has a three-point descriptive Likert-scale. Patient's answers are transformed into a scale ranging from -0.59 - 1.0 (1 equals perfect health). The change in EQ-5D from baseline to follow-up will be registered.
Time from inclusion until time for to surgery. | 10 years
A questionnaire mapping subjective change of symptoms from baseline in a 6 point response scale, ranging from completely recovered to getting worse. | Follow-up at 2,5 and 10 years
A questionnaire mapping the satisfaction with living with the current state of symptoms for the rest of the life in a 5 point response scale, ranging from very satisfied to very dissatisfied. | Follow-up at 2,5 and 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Frode G Rekeland, MD, Principal Investigator — Kysthospitalet i Hagavik, Orthopeadic clinic, Haukeland University Hospital; Clemens Weber, PhD, MD, Study Chair — Stavanger University Hospital, Department for Neurosurgery
Locations (1):
- Kysthospitalet i Hagavik, Orthopeadic clinic, Haukeland University Hospital, Hagavik, Norway

REFERENCES:
- [Derived] Indrekvam K, Myklebust TA, Austevoll IM, Hermansen E, Banitalebi H, Banerud IF, Weber C, Brisby H, Brox JI, Hellum C, Storheim K. Responsiveness of the Oswestry Disability Index and Zurich Claudication Questionnaire in patients with lumbar spinal stenosis: evaluation of surgically treated patients from the NORDSTEN study. Eur Spine J. 2024 Nov;33(11):4270-4280. doi: 10.1007/s00586-024-08440-1. Epub 2024 Aug 13. PMID 39134699
- [Derived] Indrekvam K, Banerud IF, Hermansen E, Austevoll IM, Rekeland F, Guddal MH, Solberg TK, Brox JI, Hellum C, Storheim K. The Norwegian degenerative spondylolisthesis and spinal stenosis (NORDSTEN) study: study overview, organization structure and study population. Eur Spine J. 2023 Dec;32(12):4162-4173. doi: 10.1007/s00586-023-07827-w. Epub 2023 Jul 3. PMID 37395780